CLINICAL TRIAL: NCT02315898
Title: Safety and Efficacy of Inhaled Tissue Plasminogen Activator (tPA) for the Acute Treatment of Pediatric Plastic Bronchitis
Brief Title: Inhaled Tissue Plasminogen Activator for Acute Plastic Bronchitis
Acronym: PLATyPuS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kathleen A. Stringer, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMich Inhaled tPA119678; R01FD005393 (FDA)
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Results first posted 2023-11-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Plastic Bronchitis; Protein-Losing Enteropathies; Healthy
Keywords: children, congenital heart disease, metabolomics
MeSH Terms: conditions — Protein-Losing Enteropathies; Heart Defects, Congenital | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment-inhaled tPA (Experimental): All patients with plastic bronchitis enrolled into the study will receive inhaled tPA.
  Interventions: Drug: Treatment-inhaled tPA

INTERVENTIONS:
Drug: Treatment-inhaled tPA — Enrolled patients with acute plastic bronchitis (fibrin airway casts) will receive inhaled tPA treatment. The tPA regimen will consist of 5mg every six hours for a total of 72 hours.
  Other Names: alteplase; Activase

SUMMARY:
Plastic bronchitis (PB) is a rare, most often pediatric disease characterized by the formation of obstructive airway casts primarily composed of fibrin. There is presently no FDA-approved pharmacotherapy for PB, but acute exacerbations of the illness are often treated with inhaled tissue plasminogen activator (tPA). To date, this is done somewhat anecdotally because there has been no safety or efficacy testing of this treatment. In addition, there is presently no reliable surrogate marker of adverse drug events. Nevertheless, in the absence of inhaled tPA treatment, PB-induced respiratory distress can be severe, often warranting urgent or emergent bronchoscopy for cast removal, or can sometimes result in respiratory failure. As such there is a significant unmet need for safety and efficacy testing of inhaled tPA and for biomarkers of drug response.

Objectives and Endpoints: The objectives of this protocol are to: 1) test the safety and efficacy of an inhaled tPA regimen in children with PB; and 2) identify potential candidate biomarkers of inhaled tPA drug response. Safety endpoints will consist of the development of new, active bleeding that is systemic and/or pulmonary and/or new hematuria (defined as gross hematuria). Secondary endpoints of efficacy will also be measured (e.g., frequency of cast production). Urine and blood will also be collected for the development of potential biomarkers of inhaled tPA drug response.

Funding source- FDA OOPD

DETAILED DESCRIPTION:
Background and Rationale: Plastic bronchitis (PB) is a rare, disease characterized by the formation of obstructive fibrin airway casts. Presently, acute exacerbations of the illness are often treated with inhaled tissue plasminogen activator (tPA), in part, because there are no FDA approved treatments. To date, there has been no safety or efficacy testing of inhaled tPA. In addition, there is presently no reliable marker that could be used to assess adverse drug events. However, in the absence of inhaled tPA treatment, PB-induced respiratory distress can be severe, often warranting urgent or emergent bronchoscopy for cast removal, or can sometimes result in respiratory failure. This clinical trial will address the unmet need for safety and efficacy testing of inhaled tPA and for assessing biomarkers of drug response.

Objectives and Endpoints: This is an open-label, multi-center clinical trial of inhaled tPA for the treatment of acute PB. The objectives of this protocol are to: 1) test the safety and efficacy of an inhaled tPA regimen in children with PB; and 2) identify potential candidate biomarkers of inhaled tPA drug response. Safety endpoints will consist of the development of new, active bleeding that is systemic and/or pulmonary and/or new hematuria (defined as gross hematuria). Secondary endpoints of efficacy will also be measured (e.g., frequency of cast production). Urine and blood will also be collected for the development of potential biomarkers of inhaled tPA drug response.

Assessments: Enrolled subjects will be routinely clinically monitored and blood work will be assessed for the development of new, active bleeding that is systemic and/or pulmonary or new gross hematuria. Levels of oxygenation and pulmonary function will be assessed during the study period. We will also include the incidence of expectorated casts as a measurement of efficacy.

Statistical Methods: This is an open-label study of up to 13 subjects with PB that will serve as their own controls. A group of healthy subjects (n=12), Fontan subjects without PB (n=12), and Fontan subjects with protein losing enteropathy (PLE) (n=12) will serve as controls for biomarker assay development. The incidence of new, active bleeding events and the frequency of airway cast expectoration will be assessed in subjects with PB. PLE is another illness that is associated with congenital heart disease in children that has been surgically remedied by the Fontan procedure.

The active treatment arm (inhaled tPA) will be conducted across six clinical centers. In addition, these centers will enroll PLE control patients. All other control subjects will only be enrolled at the University of Michigan.

The outcome measures only pertain to tPA treated patients. Since the control subjects are not included in the outcome analysis, recruitment/enrollment status pertains to the PB patients. The University of Michigan has initiated enrollment of healthy control subjects and there have been consented subjects.

ELIGIBILITY:
Inclusion Criteria (patients with plastic bronchitis):

1. ≥ 5 years of age but ≤24 years of age and weigh at least 18.6 kg (41 lbs).
2. Patients with CHD that have a history of PB with previous airway cast production and/or present with symptoms of an acute exacerbation (e.g., difficulty breathing, dyspnea) of PB that requires hospitalization. An acute exacerbation of PB is defined as either respiratory symptoms suspicious for airway cast formation and/or the expectoration of, or a bronchoscopy retrieved, fibrin PB cast.
3. Patients without CHD that present with an acute exacerbation of PB, defined as the expectoration of, or a bronchoscopy retrieved, fibrin PB cast that causes acute respiratory distress (e.g., severe coughing, difficulty breathing, dyspnea) or a history of PB with pathologic evidence of fibrin airway cast production. Either a cast sample (at least ½ inch (~4cm)) or a pathology report that documents PB cast fibrin content must be submitted to the UM pathology core.
4. Must be able to use a mouthpiece nebulizer.
5. Informed consent (with parental if age ≥14 years) or assent for age ≥10 and < 14 years old with parental informed consent.

Exclusion Criteria (patients with plastic bronchitis):

1. Known contraindication(s) to the use of tPA, including:

   * active internal bleeding;
   * history of cerebrovascular accident;
   * recent intracranial or intraspinal surgery or trauma;
   * intracranial neoplasm, intracranial arteriovenous malformation or intracranial aneurysm;
   * known bleeding diathesis;
   * and/or severe uncontrolled hypertension
2. Body weight >/= 100th percentile or BMI > 30
3. Known cystic fibrosis
4. Currently receiving dornase-alfa and/or inhaled unfractionated or low molecular weight heparin and/or a direct acting oral anticoagulant (e.g., dabigatran, rivaroxaban)

   * Inhaled unfractionated or low molecular weight heparin must be discontinued at least 72h. Inhaled dornase alfa should be discontinued no later than the time of the start of enrollment in the treatment phase. If the patient is receiving inhaled tPA, this regimen must be discontinued and transitioned to the inpatient dosing regimen (5mg Q6h) of study drug.
   * Direct acting oral anticoagulants must be discontinued one week prior to the start of enrollment in the treatment phase.
5. Protein losing enteropathy
6. Liver dysfunction (defined as ≥ 3X the normal levels of one or both liver transaminases, AST and AST)

   • Transaminase levels acquired within the last 9 months can be used to assess liver function. If previously normal and there is no clinical indication that liver function has worsened, the patient can be enrolled. If there are no transaminase values within the last 9 months, they need to be acquired as part of screening
7. Need for concomitant intravenous or sub-cutaneous anti-coagulation with resulting anti- Xa levels > 0.5 (low molecular weight heparins) or > 0.3 (unfractionated heparin)
8. International normalized ratio (INR) > 2.0 if not receiving warfarin
9. Patients being actively treated for thrombosis
10. Concomitant use of a thienopyridine class antiplatelet agent (e.g., clopidogrel)
11. A platelet count of < 100,000 platelets/µL
12. A hematocrit <30%
13. Gross hematuria on screening urinalysis
14. Pregnant or lactating women (negative pregnancy test required for girls/women of childbearing potential at the time of inhaled tPA administration). All women of child- bearing potential must be willing to practice appropriate contraception throughout the study.
15. Subjects who are known positive for, or are hospitalized with COVID-19 caused by the new coronavirus, SARS CoV-2, at the start of the treatment phase.
16. Suspected or active concurrent infectious illness.

Inclusion Criteria for Healthy Controls

1. Healthy children ≥ 5 years of age but ≤18 years of age with no other underlying concomitant illness or chronic medication use (with the exception of vitamin supplements)
2. Weigh at least 18.6 kg (41 lbs)

Inclusion Criteria for Healthy non-PB Fontan Controls

1. Children ≥ 5 years of age but ≤18 years of age with uncomplicated Fontan physiology with no history of PB, other Fontan-associated complications (e.g., hepatopathy, PLE), or other concomitant illnesses (e.g., asthma).
2. Weigh at least 18.6 kg (41 lbs)

Inclusion Criteria for PLE Fontan Controls

1. Children ≥ 5 years of age but ≤18 years of age with Fontan physiology, no history of PB and a diagnosis of PLE defined as clinically symptomatic hypoproteinemia and/or enteral protein loss.
2. Weigh at least 18.6 kg (41 lbs)

Exclusion Criteria for Healthy, non-PB Fontan Controls and PLE Fontan Controls

1. Exceed the 100th percentile for body weight or have a BMI greater than 30.
2. History of post-operative chylothorax following any palliation surgery (except for PLE controls).
3. Known liver dysfunction per medical record review (e.g., defined as ≥ 3X the normal levels of one or both liver transaminases [ALT & AST])
4. COVID-19 positive within the last 14 days prior to the scheduled visit and/or the presence of symptoms consistent with COVID-19 at the time of the visit
5. Suspected or active concurrent infectious illness

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Stringer, PharmD, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital, Stanford University, Palo Alto, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan Mott Children's Hospital, Ann Arbor, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Caroline, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared in accordance with the NIH's policy on data sharing. The University of Michigan has options for data repository (e.g., ICPSR, http://www.icpsr.umich.edu/icpsrweb/deposit/). All metabolomics data will be deposited in the NIH's Metabolomics Workbench (http://www.metabolomicsworkbench.org/). The study PI will also honor requests made by individual investigators.

REFERENCES:
- [Derived] Stringer KA, Goldberg D, Chen S, Thrush P, Graham EM, Lubert A, Myers J, McLellan L, Flott T, Nasr S, Schumacher KR. A Multicenter, Open-Label Study to Assess the Safety of Nebulized Tissue Plasminogen Activator for the Acute Treatment of Pediatric Plastic Bronchitis: The PLATyPuS Trial. Pharmacotherapy. 2025 Oct;45(10):677-687. doi: 10.1002/phar.70056. Epub 2025 Sep 5. PMID 40910281

RESULTS

PARTICIPANT FLOW:
Groups:
- PLE Controls: Participants with congenital heart disease and protein losing enteropathy but with no history of plastic bronchitis
- Fontan Controls: Participants with Fontan physiology with no history of plastic bronchitis or PLE
- Healthy Controls: Participants without congenital heart disease and no history of pulmonary disease (including plastic bronchitis) or protein losing enteropathy
Period: Overall Study
Arm/Group | Treatment-inhaled tPA | PLE Controls | Fontan Controls | Healthy Controls
Started | 10 | 8 | 9 | 13
Completed | 8 | 8 | 9 | 12
Not Completed | 2 | 0 | 0 | 1
Not completed — 2 in the treatment arm did not meet treatment eligibility; a healthy control screen failed | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-inhaled tPA | PLE Controls | Fontan Controls | Healthy Controls | Total
Number analyzed (Participants) | 8 | 8 | 9 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean (SD) age in years Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
  years | 12.1 (4.1) | 13 (2.6) | 14 (3.2) | 11.7 (2.5) | 12.6 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
  Participants
    sex: Female | 4 | 1 | 4 | 4 | 13
    sex: Male | 4 | 7 | 5 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
  Participants
    Hispanic or Latino | 2 | 2 | 0 | 2 | 6
    Not Hispanic or Latino | 6 | 6 | 9 | 7 | 28
    Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 0 | 0 | 2
    White | 5 | 4 | 8 | 11 | 28
    More than one race | 2 | 3 | 0 | 0 | 5
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: Two participants in the Treatment arm were enrolled but were not treated because they did not have a subsequent episode of acute plastic bronchitis. One healthy control participant was enrolled and did not complete the study due to a screen failure.
  participants
    United States | 8 | 8 | 9 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Number of Subjects That Develop New, Active Bleeding
Description: The number of subjects with new systemic and/or pulmonary and/or gross hematuria
Time Frame: Participants will be assessed every 24 hours (daily) for the duration of tPA treatment which was up to 4 days and at hospital discharge which typically occurred within 1 week of treatment initiation.
Population: The number of new, active systemic bleeding events were assessed for participants enrolled in the treatment arm only. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Participants | 0

2. Secondary Outcome: Arterial Oxygen Saturation (%)
Description: Changes in oxygen saturation (%) will be monitored by pulse oximetry (oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin in the blood). Since this measurement was made at different times for each participant, the mean (SD) oxygen saturation (%) prior to study drug administration (pre-treatment) and at hospital discharge (~ 1 week post-treatment) was calculated.
Time Frame: Participants will be assessed at screening (if applicable), just prior to treatment and daily for the duration of tPA treatment, up to 4 days, at hospital discharge (~ 1 week) and again at 30 days.
Population: Oxygen saturation was assessed at screening (if applicable), prior to treatment and daily for the duration of tPA treatment, at hospital discharged and at 30 days. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
  Because pulse oximetry was measured at different times during hospitalization across patients, we report the mean pre-treatment and the hospital discharge (~1 week post-treatment) mean (SD) values.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
percent
  Pre-treatment | 90.6 (4.7)
  Post-treatment (hospital discharge): number analyzed (Participants) | 7
  Post-treatment (hospital discharge) | 90.6 (4.2)

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: The change in FEV1 (L) from pre- to post- tPA treatment will be assessed for each patient.
Time Frame: Participants will be assessed at screening (if applicable), just prior to treatment and then daily for the duration of tPA treatment, up to 4 days, at hospital discharge and again at 30 days.
Population: The FEV1 (L) was assessed prior to and during inhaled tPA treatment, at hospital discharge and at the 30 d follow up visit. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
  Many treatment arm participants did not have values at all time points.The outcome measure is the pre-treatment average, the overall average during treatment (days 0-4) and the average at hospital discharge (~ 1 week) after treatment initiation.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Liters
  Pre-treatment: number analyzed (Participants) | 3
  Pre-treatment | 1.7 (0.95)
  Treatment (days 0-4): number analyzed (Participants) | 7
  Treatment (days 0-4) | 1.60 (0.62)
  Hospital Discharge (~1 week): number analyzed (Participants) | 5
  Hospital Discharge (~1 week) | 1.42 (0.66)

4. Secondary Outcome: Forced Expiratory Flow 25-75% (FEF25-75)
Description: The FEF25-75 will be assessed for each patient in the treatment arm prior to study drug, during study drug administration (days 0-4), at hospital discharge (~ 1 week after treatment) and again at 30 days.
Time Frame: as for outcome 3
Population: The FEF25-75 will be assessed for each patient in the treatment arm. This is because the outcome measures were per-specified to collect data only from the treatment-inhaled tPA arm of the study.
  Many treatment arm participants did not have values at all time points.The outcome measure is the pre-treatment average, the overall average during treatment (days 0-4) and the average at hospital discharge (~ 1 week) after treatment initiation.
Measure: Mean (Standard Deviation); unit: Liters/second
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Liters/second
  Pre-treatment: number analyzed (Participants) | 2
  Pre-treatment | 1.23 (0.2)
  Treatment (days 0-4): number analyzed (Participants) | 7
  Treatment (days 0-4) | 1.76 (0.94)
  Hospital discharge (~1 week): number analyzed (Participants) | 4
  Hospital discharge (~1 week) | 1.14 (0.09)

5. Secondary Outcome: Forced Vital Capacity (FVC)
Description: The FVC (L) from prior to, during and after tPA treatment will be assessed for each patient.
Time Frame: as for outcome 3
Population: The FVC (L) before, during and after tPA treatment will be assessed. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
  Many treatment arm participants did not have values at all time points.The outcome measure is the pre-treatment average, the overall average during treatment (days 0-4) and the average at hospital discharge (~ 1 week) after treatment initiation.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Liters
  Pre-treatment: number analyzed (Participants) | 3
  Pre-treatment | 2.0 (1.14)
  Treatment (days 0-4): number analyzed (Participants) | 7
  Treatment (days 0-4) | 1.91 (0.66)
  Hospital discharge (~1 week): number analyzed (Participants) | 5
  Hospital discharge (~1 week) | 1.80 (0.65)

6. Secondary Outcome: Frequency of Production/Expectoration of Airway Casts
Description: Episodes of the production of airway casts by participants enrolled in the treatment arm will be assessed.
Time Frame: Episodes of cast production will be assessed daily for the duration tPA treatment, up to 4 days and from hospital discharge (~1 week after treatment) up to 30 days
Population: Assessment of cast production during the study period was made in the PB treatment arm only. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study. This was based on self report. Cast sizes were not assessed or reported.
  The cumulative number of episodes of cast production reported at 30 days is reported.
Measure: Number; unit: episodes of cast production (30d)
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
episodes of cast production (30d) | 9

7. Secondary Outcome: Changes in the Chest X-ray (CXR)
Description: tPA treatment-induced changes in the CXR will be assessed. The chest x-ray will be scored prior to and after tPA treatment at hospital discharge (~1 week post treatment). The scores will be derived using the Brasfield scoring system which assesses air trapping, linear markings (bronchial wall thickness), bronchiectasis, lobar involvement and overall severity. A score of 25 represents a normal CXR. Points are deducted from 25 for abnormalities so the lower the score the greater the disease severity.
Time Frame: A CXR will be acquired and assessed two times during the study- once just prior to the initiation of study drug and again at hospital discharge, up to ~1 week.
Population: All patients that received tPA. CXRs were scored by a pediatric pulmonologist using the Brasfield scoring system. A score of 25 represents a normal CXR. Points are deducted from 25 for abnormalities so the lower the score the greater the disease severity. This outcome was pre-specified for the treatment arm of the study only; CXRs were not obtained in the control arms.
Measure: Mean (Standard Deviation); unit: score on a scale (0-25 normal)
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
score on a scale (0-25 normal)
  Pre-treatment | 20.6 (0.74)
  Post-treatment: number analyzed (Participants) | 7
  Post-treatment | 20.9 (0.90)

8. Secondary Outcome: Requirement for Urgent or Emergent Bronchoscopy
Description: Requirement for urgent or emergent bronchoscopy during treatment was assessed.
Time Frame: Participants will be followed for the duration of tPA treatment, up to 4 days.
Population: The number of treatment arm participants who required urgent or emergent bronchoscopy was recorded. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Participants | 0

9. Secondary Outcome: Requirement for Mechanical Ventilation
Description: Requirement for mechanical ventilation will be assessed in participants enrolled in the treatment arm during the treatment period.
Time Frame: Participants will be followed for the duration of tPA treatment, up to 4 days.
Population: The number of participants in the treatment arm who required mechanical ventilation was recorded. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
Participants | 0

10. Secondary Outcome: Pathological Assessment (Qualitative) of Fibrin and Mucin Content of Airway Casts
Description: PB cast fibrin and mucin content will be qualitatively assessed in casts that are collected before and after tPA treatment up to hospital discharge (~1 week) by a co-investigator pathologist. Each cast will be qualitatively assessed for fibrin and mucin content based on standard pathological procedures.
Time Frame: Available (submitted) airway casts will assessed for the duration of the hospital stay, up to hospital discharge (~1 week).
Population: Any PB casts that were expectorated by treatment participants were sent for pathological analysis of casts by UM pathology. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study.
  None of the PB-tPA treated study participants produced and submitted airway casts for pathological assessment. Therefore, no data are available for this outcome measure.
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 0

11. Secondary Outcome: Detection of Fibrin Degradation Product (FDP) in the Systemic Circulation
Description: Blood samples will be assayed for FDP (mg/L) during the study. This is a measure of fibrin degradation in the blood and is a value that can be altered by tPA treatment. An FDP (or D-dimer) value <0.5 mg/L is considered normal.
Time Frame: FDP will be assessed at screening (if applicable), prior to treatment and then daily during the hospital stay (~1 week) and again at 30 days
Population: Blood levels of FDP were assessed from participants in the treatment arm of the study. This is because the outcome measures were pre-specified to collect data only from the treatment-inhaled tPA arm of the study. The pre-treatment average of participants and the post-treatment average (at hospital discharge, ~ 1 week from the start of treatment) are reported.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 8
mg/L
  Pre-treatment: number analyzed (Participants) | 5
  Pre-treatment | 0.32 (0.08)
  Hospital discharge (~1 week): number analyzed (Participants) | 5
  Hospital discharge (~1 week) | 4.14 (4.11)

12. Secondary Outcome: Assessment of Patient Centered Outcomes
Description: We will use a questionnaire to assess how many participants had changes in quality of life related to plastic bronchitis and its treatment during the study in participants enrolled in the treatment arm. For this, the Cystic Fibrosis Questionnaire-Revised (CFQ-R) will be used since there is not a specific plastic bronchitis questionnaire. The CFQ-R is designed to measure impact on overall health, daily life, perceived well-being and symptoms. The CFQ-R uses a Likert scale to rate nine quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions and three symptom scales: Weight, respiratory, and digestion. Each item is summed to generate a domain score. Scores range from 0 to 100, with higher scores indicating better health.
Time Frame: This measurement will be performed prior to tPA treatment, at hospital discharge (~ 1 week) and again at 30 days.
Population: The number of participants enrolled in the treatment arm who had a relevant change in CTQ-R questionnaire domain scores from pre-treatment to hospital discharge were not able to be assessed because there were no participants who completed questionnaires at these two time points. No data are available for this secondary outcome.
Arm/Group | Treatment-inhaled tPA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: For the treatment arm of the study, AEs were systematic assessed during hospitalization and tPA treatment (measurements and routine clinical assessments for bleeding). Following hospital discharge, adverse events information collection was non-systematic, self-reporting.
  For the control participants, AEs were assessed at time of their one time study visit. These participants did not receive study drug.
Arm/Group | Treatment-inhaled tPA | PLE Controls | Fontan Controls | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 8/8 | 0/8 | 0/9 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-inhaled tPA (N=8) | PLE Controls (N=8) | Fontan Controls (N=9) | Healthy Controls (N=12)
serious adverse event (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — A patient received a heart transplant during the study period. This was not a study-drug related event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-inhaled tPA (N=8) | PLE Controls (N=8) | Fontan Controls (N=9) | Healthy Controls (N=12)
blood-tinged mucus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
coughing (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
nose bleed (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
vasovagal response to venipuncture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor appetite and constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile to 39.1 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythematous and congested throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased pleural effusion on chest x-ray (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patchy lobe atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal labs on day 30 IgG, D-dimer (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated D-dimer (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated WBC count (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a small (n=8) safety trial of inhaled tPA in pediatric patients with the extraordinarily rare disease, plastic bronchitis. As such, no statistical analysis can confidently be performed so the findings are descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT02315898/Prot_SAP_000.pdf